CLINICAL TRIAL: NCT06769724
Title: Anthropometric Predictability of Full-Thickness Peroneus Longus and Semitendinosus Autograft Size: A Comparative Analysis
Brief Title: Anthropometric Predictability of Full-Thickness Peroneus Longus and Semitendinosus Autograft Size
Status: Recruiting | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Fevzi Gurkan Aslan, Dr, Karadeniz Technical University
Other Study IDs: 24237859611
Record Dates: First submitted 2025-01-01; First posted 2025-01-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligaments
Keywords: Anterior Cruciate Ligaments; peroneus longus tendon; semitendinosus tendon; anthropometric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Semitendinosus Tendon: The participiants underwent acl reconstruction with semitendinosus tendon autograft
  Interventions: Procedure: Anterior cruciate ligament reconstruction surgery
- Peroneus Longus Tendon: The participiants underwent acl reconstruction with peroneus longus tendon autograft
  Interventions: Procedure: Anterior cruciate ligament reconstruction surgery

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction surgery — Anterior cruciate ligament reconstruction surgery with semitendinosus tendon autograft
  Groups: Semitendinosus Tendon
Procedure: Anterior cruciate ligament reconstruction surgery — Anterior cruciate ligament reconstruction surgery with peroneus longus autograft
  Groups: Peroneus Longus Tendon

SUMMARY:
The study is aimed to determine correlation between autografts used in anterior cruciate ligaments and anthropometric variables e.g. height, sex, weight, BMI etc..

DETAILED DESCRIPTION:
Categorical data: Age, Sex, Height, Weight, BMI, Preoperative parameters: cruris length, cruris circumference, thigh length, thigh circumference Intraoperative Info: Tendon Type, Tendon length (total-muscular part-tendinoz part), Graft Length, Graft Diameter.

After the data collected, correlation analysis will be held and determine the both tendons preoperative size predictability before acl reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-45 years
* Diagnosed Acl rupture preoperavitely with mri imaging
* Diagnosed Acl rupture and having symptoms related to acl rupture
* Eligible for harvesting same side semitendinosus or peroneous longus tendon

Exclusion Criteria:

* Previous surgery history on donor side knee or ankle
* Congenital defect on donor extremity
* Multiple Ligament Injury History

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who will apply to our center due to ACL ligament injury and will be decided to undergo surgical treatment will be included in the study if they volunteer to participate.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Preoperative Anthropometric Variables and Autograft Dimensions | Intraoperatively
  To assess the correlation between preoperative anthropometric measurements and intraoperative autograft dimensions

SECONDARY OUTCOMES:
Comparison of Predictability Between Peroneus Longus and Semitendinosus Tendons | Preoperatively at surgery day
  To determine whether the predictability of tendon dimensions based on anthropometric variables,height(cm), weight(kg), BMI(kg/m^2), cruris length(cm), and circumference(cm) for estimating tendon and graft size before surgery, differs between peroneus longus and semitendinosus autografts.
Predictability of Autograft Dimensions Based on Preoperative Anthropometric Data | Intraoperatively
  To evaluate the predictive power of anthropometric variables (height(cm), weight(kg), BMI(kg/m^2), cruris length(cm), and circumference(cm)) for estimating tendon and graft size(cm) before surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Orthopedic and Traumatology Department, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Wierer G, Gwinner C, Scheffler S. Peroneus Longus Split Versus Semitendinosus Tendon Autograft Size: A Cross-sectional Study. Am J Sports Med. 2023 Jun;51(7):1743-1751. doi: 10.1177/03635465231165297. Epub 2023 Apr 24. PMID 37092720